CLINICAL TRIAL: NCT02622971
Title: Isolated and Combined Effects of Phototherapy and Cryotherapy in Post-exercise Skeletal Muscle Recovery
Brief Title: Phototherapy and Cryotherapy in Post-exercise Skeletal Muscle Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Collaborators: Multi Radiance Medical (Industry)
Responsible Party: Principal Investigator, Adriane Aver Vanin, PhD candidate, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CEP 470.174
Record Dates: First submitted 2015-11-24; First posted 2015-12-07 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Post-exercise Muscle Recovery
Keywords: phototherapy; cryotherapy; exercise; fatigue; recovery
MeSH Terms: conditions — Motor Activity; Fatigue | interventions — Low-Level Light Therapy; Cryotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- PBMT and Cryotherapy (Active Comparator): Volunteers allocated in this group received phototherapy (PBMT - applied in six points of quadriceps) and cryotherapy (20 minutes in PRICE protocol) as a treatment three minutes and 24h, 48h and 72h after exercise protocol.
  Interventions: Other: PBMT; Other: Cryotherapy
- Cryotherapy and PBMT (Active Comparator): Volunteers allocated in this group received cryotherapy (20 minutes in PRICE protocol) and phototherapy (PBMT - applied in six points of quadriceps) as a treatment three minutes and 24h, 48h and 72h after exercise protocol.
  Interventions: Other: PBMT; Other: Cryotherapy
- PBMT (active phototherapy) (Active Comparator): Volunteers allocated in this group received active phototherapy (PBMT - applied in six points of quadriceps) as a treatment three minutes and 24h, 48h and 72h after exercise protocol.
  Interventions: Other: PBMT
- PBMT (placebo phototherapy) (Placebo Comparator): Volunteers allocated in this group received placebo phototherapy (PBMT - applied in six points of quadriceps) as a treatment three minutes and 24h, 48h and 72h after exercise protocol. The placebo PBMT device was identical to the active devices and displayed the same settings and emitted the same sound regardless of the comparator.
  Interventions: Other: PBMT
- Cryotherapy (Active Comparator): Volunteers allocated in this group cryotherapy (20 minutes in PRICE protocol) as a treatment three minutes and 24h, 48h and 72h after exercise protocol. Two flexible ice packs filled with ice cubes and water (with a volume of 1.15 liters each) were used in order to cover the entire quadriceps. Rubber belts were used to apply compression and to affix the packs tightly to the volunteers' quadriceps.
  Interventions: Other: Cryotherapy

INTERVENTIONS:
Other: PBMT — Effects of phototherapy isolated and/or combined with cryotherapy in post-exercise skeletal muscle recovery.
  Other Names: photobiomodulation therapy
  Arms: Cryotherapy and PBMT; PBMT (active phototherapy); PBMT (placebo phototherapy); PBMT and Cryotherapy
Other: Cryotherapy — Effects of cryotherapy isolated and/or combined with phototherapy in post-exercise skeletal muscle recovery.
  Arms: Cryotherapy; Cryotherapy and PBMT; PBMT and Cryotherapy

SUMMARY:
Volunteers were divided randomly in five experimental groups. VAS (Visual Analogic scale) to measure DOMS (Delayed Onset Muscle Soreness) and blood samples was taken before any procedure. Then, volunteers performed stretching and warm-up followed by MVC test (isometric test in isokinetic dynamometer to measure muscle function). After, volunteers performed the exercise protocol (75 eccentric contractions) to lead to muscle fatigue. Immediately after exercise protocol (1 minute) and 1 hour, 24, 48, 72 and 96 hours after, blood sample, VAS measure and MVC test were repeated. The treatments according to randomisation were performed three minutes after exercise protocol and it were performed again in 24, 48, 72h after eccentric exercise.

The variables regarding to muscle function (MVC, DOMS) and the indirect marker of muscle damage (CK activity) were monitored in all time points mentioned above (baseline, 1 minute, 1 hour, 24, 48, 72 and 96 hours after exercise protocol).

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled clinical trial was performed at the Laboratory of Phototherapy in Sport and Exercise at Nove de Julho University in the city of São Paulo, Brazil.

Fifty healthy untrained male subjects were recruited from university staff and students to participate in the study. All participants voluntarily must agree to participate and they signed the informed consent statement. The intention-to-treat analysis was followed.

The volunteers were randomly allocated to five experimental groups (n=10 per group) according to the applied comparator. Randomisation was carried out by a simple drawing of lots (A, B, C, D or E). Blood samples (10 ml) was taken by a qualified nurse to analyse CK activity posteriorly. This blood collection was repeated 1 minute, 1 hour, 24, 48, 72 and 96 hours after eccentric protocol.

A visual analogue scale (VAS) of 100 mm was used as a self-rating of volunteers DOMS intensity, with assistance of a blinded researcher. DOMS assessments were performed at baseline, immediately after eccentric exercise protocol (1 minute), and it was repeated at 1, 24, 48, 72 and 96 hours after the exercise protocol. Before exercise protocol, volunteers will perform a stretching and warm-up of the non-dominant lower limb and then they will perform Maximum voluntary contraction (MVC) to evaluate muscle function. MVC measurements were repeated at the same time intervals as the CK measures.

The exercise protocol consists in 75 eccentric isokinetic contractions of the knee extensor musculature in the non-dominant leg (5 sets of 15 repetitions, 30-second rest interval between sets) at a velocity of 60°.seg-1 in both the eccentric and concentric movements with a 60° range of motion (between 90° and 30° of knee flexion).

Regarding to treatment, all volunteers received the treatment according to randomisation three minutes after eccentric exercise protocol. Comparators were repeated at 24, 48, and 72 hours following the collection of additional blood samples for CK analyses and MVC and DOMS assessments.

The five groups was divided in: PBMT (photobiomodulation therapy)+cryotherapy; cryotherapy+PBMT; active PBMT; placebo PBMT and only cryotherapy.

PBMT was applied employing a cordless, portable GameDay™ Super Pulsed Laser (manufactured by Multi Radiance Medical, USA) to 6 sites of quadriceps femoris in direct contact with the skin (2 centrally - rectus femoral and vastus intermedius; 2 laterally - vastus lateralis; and 2 medially - vastus medialis) and cryotherapy was done with two flexible ice packs filled with ice cubes and water (with a volume of 1.15 liters each) that will cover the entire quadriceps for 20 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Subjects were included in the study if they performed less than 2 exercise session per week

Exclusion Criteria:

* Subjects were excluded if occurred any musculoskeletal injury to hips or knees within the previous two months,
* if they were currently using pharmacological agents or nutritional supplements regularly,
* if a musculoskeletal injury during the study occurred or if they reported use of either alcohol or tobacco.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2014-06; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Maximum voluntary contraction (MVC) | one week
  The MVC test consisted of three five-second isometric contractions of the knee extensors of the non-dominant leg. The highest torque value of the three contractions (peak torque) was used for statistical analysis.

SECONDARY OUTCOMES:
Evaluation of Delayed Onset Muscle Soreness (DOMS) | one week
  A visual analogue scale (VAS) of 100 mm was used as a self-rating of volunteers DOMS intensity, with assistance of a blinded researcher.
CK (Creatine Kinase) activity | one week
  Blood samples (10 ml) was taken by a qualified nurse blinded to the allocation of the volunteers to the five experimental groups from the antecubital vein. Spectrophotometry and specific reagent kits (Labtest®, São Paulo - SP, Brazil) were used to analyze CK (Creatine Kinase) activity as an indirect marker of muscle damage.

CONTACTS AND LOCATIONS:
Overall Officials: Ernesto Cesar P Leal-Junior, PhD, PT, Principal Investigator — University of Nove de Julho
Locations (1):
- Laboratory of Phototherapy in Sports and Exercise, Universidade Nove de Julho (UNINOVE), São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
all data is stored and saved in electronic devices to clarify any possible doubt regarding to methodological procedures and results.

REFERENCES:
- [Result] Antonialli FC, De Marchi T, Tomazoni SS, Vanin AA, dos Santos Grandinetti V, de Paiva PR, Pinto HD, Miranda EF, de Tarso Camillo de Carvalho P, Leal-Junior EC. Phototherapy in skeletal muscle performance and recovery after exercise: effect of combination of super-pulsed laser and light-emitting diodes. Lasers Med Sci. 2014 Nov;29(6):1967-76. doi: 10.1007/s10103-014-1611-7. Epub 2014 Jun 19. PMID 24942380
- [Result] Grandinetti Vdos S, Miranda EF, Johnson DS, de Paiva PR, Tomazoni SS, Vanin AA, Albuquerque-Pontes GM, Frigo L, Marcos RL, de Carvalho Pde T, Leal-Junior EC. The thermal impact of phototherapy with concurrent super-pulsed lasers and red and infrared LEDs on human skin. Lasers Med Sci. 2015 Jul;30(5):1575-81. doi: 10.1007/s10103-015-1755-0. Epub 2015 May 19. PMID 25987340
- [Result] Baroni BM, Leal Junior EC, De Marchi T, Lopes AL, Salvador M, Vaz MA. Low level laser therapy before eccentric exercise reduces muscle damage markers in humans. Eur J Appl Physiol. 2010 Nov;110(4):789-96. doi: 10.1007/s00421-010-1562-z. Epub 2010 Jul 3. PMID 20602109
- [Result] Graham CA, Stevenson J. Frozen chips: an unusual cause of severe frostbite injury. Br J Sports Med. 2000 Oct;34(5):382-3. doi: 10.1136/bjsm.34.5.382. PMID 11049150
- [Result] Moeller JL, Monroe J, McKeag DB. Cryotherapy-induced common peroneal nerve palsy. Clin J Sport Med. 1997 Jul;7(3):212-6. doi: 10.1097/00042752-199707000-00011. PMID 9262890
- [Result] Bassett FH 3rd, Kirkpatrick JS, Engelhardt DL, Malone TR. Cryotherapy-induced nerve injury. Am J Sports Med. 1992 Sep-Oct;20(5):516-8. doi: 10.1177/036354659202000505. PMID 1443317